CLINICAL TRIAL: NCT07034859
Title: Cabergoline in the Management of Nonfunctioning Pituitary Adenoma
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Beihu Branch (Other); National Taiwan University (Other); National Taiwan University Hospital Hsin-Chu Branch (Other); National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301198MINB
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pituitary Adenoma; MRI; RCT
Keywords: cabergoline; nonfunctioning pituitary adenoma; randomized controlled trial
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving cabergoline treatment (Experimental): Cabergoline (Dostinex ®) 0.5 mg/tablet. Cabergoline will be given orally 1mg/week (Day1-14), 2mg/week (Day15-end of the study).
  Interventions: Drug: Cabergoline 0.5 MG
- Control (No Intervention): Participants without carbergoline treatment

INTERVENTIONS:
Drug: Cabergoline 0.5 MG — Cabergoline (Dostinex ®) 0.5 mg/tablet. Cabergoline will be given orally 1mg/week (Day1-14), 2mg/week (Day15-end of the study).
  Arms: Participants receiving cabergoline treatment

SUMMARY:
The goal of this clinical trial is to learn if Cabergoline (Dostinex), a dopamine agonist which has been widely used to treat hyperprolactinemia, prolactinoma for many years, works to treat nonfunctioning pituitary adenoma (NFPA) in adults. The main questions it aims to answer are:

Does cabergoline reduce the size of NFPA effectively when used as primary therapy?

Participants will:

Be 1:1 randomized into two groups. Either to take cabergoline or none for 48 weeks, Visit the clinic every 12 weeks for checkups and tests, Undergo scheduled imaging studies, Magnetic Resonance Imaging (MRI) to measure the change of tumor size.

DETAILED DESCRIPTION:
1. BACKGROUND and study rationale The overall prevalence of pituitary adenoma in the general population ranges from 1 in 865 to 1 in 2688 adults. Of these tumors, between 15% and 54% are nonfunctioning pituitary adenomas (NFPAs). Most NFPAs are macroadenomas with diameter greater than 10 mm. Generally, surgery is recommended as first-line treatment of symptomatic NFPAs. However, medical therapies or radiation therapy or active surveillance may be indicated for some patients.

   Cabergoline (Dostinex), a dopamine agonist which has been widely used to treat hyperprolactinemia, prolactinoma for many years. For NFPA, there were studies revealing that dopamine agonists might reduce residual tumor size postoperatively. But those studies were most observational studies and performed retrospectively. There is only one randomized controlled trial assessing the effect of cabergoline on post-operative residual NFPA. The result showed cabergoline was an effective drug for treating residual NFPA, and its use was associated with a high rate of tumor shrinkage. Therefore, nowadays dopamine agonist treatment is usually reserved for the treatment of residual tumor postoperatively. Though, there were reports showing dopamine agonist may reduce the size of NFPAs. Nevertheless, there is no report using dopamine agonist as primary treatment of NFPAs, especially preoperatively.

   Furthermore, responsible mechanisms of dopamine agonists in NFPA remain poorly understood. Therefore, randomized controlled trial focusing on the effect of dopamine agonists on NFPA is needed.

   Hence, we designed a multicenter, open-label, randomized, controlled parallel study to evaluate the effect of cabergoline on the tumor size among patients diagnosed with NFPA.
2. STUDY OBJECTIVES 2.1 Primary Objective The primary objective is to assess the effect of cabergoline on tumor size by comparing the proportion of tumor shrinkage between cabergoline and control group. The change of tumor size will be measured by the maximal diameter of tumor and estimated volume of the tumor over the 48 week-treatment period.

   2.2 Secondary Objectives The secondary objective is to assess the effect of cabergoline via measurement of progression -free survival (PFS) over the 48 week-treatment period. Besides, the largest diameter of tumor and estimated volume of tumor will also be recorded and compared between groups.
3. STUDY DESIGN 3.1 Study Overview This is a multiple center, open-labeled, controlled, randomized, parallel study. 30 of subjects over 18 years old are planned. Subjects must be consenting adult volunteers who were diagnosed with NFPA, whose tumor size are at least 0.5cm in diameter and recent serum prolactin levels are less than 30ng/ml. Besides, subjects used to undergo either brain surgery or radiotherapy, subjects currently receiving any product of dopamine agonist will not be enrolled.

   Subjects will be 1:1 randomized to treatment group or controlled group. Each subject will be administered with added-on either cabergoline (treatment group) or none (control group) for total 48 weeks. In treatment group, cabergoline 0.5mg/tablet will be given from 1mg per week (1 tab BIW) for 2 weeks (Day1~14), then titrate up to 2mg per week (2 tabs BIW) since Day 15 till end of the study. The subjects will come for 7 visits during the study. Visit 1 and 2 must occur within 14 days of each other, visit 3 will be 2 weeks after visit 2, visit 4 will be 10 weeks after visit 3, all the rest visits will be 12 weeks (± 3days) apart. Volunteers will be screened at visit 1, and if they meet the inclusion/exclusion criteria, they will be entered into the study and randomized into 2 groups for inclusion at visit 2.

   Ideally, the following treatment regimens will be used:

   Group A: Cabergoline orally 1mg/week (Day1-14), 2mg/week (Day15-end of the study) Group B: None Total duration of subject participation will be 50 weeks. Total duration of the study is expected to be 5 years (Enrollment to final data analysis).
4. Criteria for evaluation 4.1 Primary Efficacy Endpoint

   * Proportion of tumor shrinkage (visit 4, 5, 7) 4.2 Secondary Efficacy Endpoints
   * Progression-free survival (visit 4, 5, 7)
   * Volume of tumor (visit 4, 5, 7)
   * Largest diameter of tumor (visit 4, 5, 7)

   4.3 Safety Evaluations
   * Incidence of cardiac valvar alteration
   * Incidence of adverse events
5. SUBJECT SELECTION 5.1 Study Population Subjects with a diagnosis of NFPA who meet the inclusion and exclusion criteria will be eligible for participation in this study.

5.2 Inclusion Criteria

1. Male ≥ 18 years of age at Visit 1
2. Documentation of NFPA as evidenced by one or more of the following criteria:

   1. Tumor size ≥ 0.5 cm in diameter.
   2. Serum prolactin level ≤ 30 ng/ml
3. Absence of previous radiotherapy or radiosurgery.
4. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

5.3 Exclusion Criteria

1. Allergic to cabergoline or ergotamine
2. Currently receiving cabergoline
3. With moderate to severe symptoms of mass effect, such as visual defect, headache, cranial nerve palsy.
4. AST, ALT over 2.5 times of the upper limit.
5. Chronic kidney disease, stage 4 and 5.
6. Hypotension
7. History of congestive heart failure, NYHA Fc III, IV
8. History of moderate or severe valvular heart disease.
9. History of Parkinson's disease.
10. History of pulmonary fibrosis
11. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
12. History of previous pituitary surgery or radiotherapy
13. Psychotic psychiatric disease
14. Active gastrointestinal tract bleeding
15. History of Raynaud's phenomenon Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

6 Concurrent Medications All subjects should be maintained on the same medications throughout the entire study period, as medically feasible, with no introduction of new chronic therapies.

6.1 Prohibited Medications and Treatments The following medications are prohibited during the study and administration will be considered a protocol violation.

* Prohibited:

  * Metoclopramide
  * Phenothiazines
  * Butyrophenones
  * Thioxanthenes
* With caution:

  * Anti-Hypertensives
  * Ergotamine

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at Visit 1.
* Documentation of NFPA as evidenced by diagnostic criteria and size ≥ 0.5 cm in diameter.
* Absence of previous hormonal pituitary hypersecretion, except prolactin level ≤ 30 ng/ml
* Absence of previous radiotherapy or radiosurgery
* Written informed consent

Exclusion Criteria:

* Allergic to cabergoline or ergotamine
* Currently receiving cabergoline
* With moderate to severe symptoms of mass effect, such as visual defect, headache, cranial nerve palsy.
* AST, ALT over 2.5 times of the upper limit.
* Chronic kidney disease, stage 4 and 5.
* Hypotension
* History of congestive heart failure, NYHA Fc III, IV
* History of moderate or severe valvular heart disease.
* History of Parkinson's disease.
* History of pulmonary fibrosis
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* History of previous pituitary surgery or radiotherapy
* Psychotic psychiatric disease
* Active gastrointestinal tract bleeding
* History of Raynaud's phenomenon
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportions of tumor shrinkage after 48 week-treatment | Baseline (Visit 1), 12th Week (Visit 4), 24th Week (Visit 5), 48th Week (Visit 7)
  The tumor volume will be calculated via ITK-SNAP version 3.6.0 at visit 1, 4, 5, 7. The largest diameter of tumor will also be measured at visit 1, 4, 5, 7. The within-group differences were examined by Wilcoxon signed-rank test. The between-group differences were examined by Wilcoxon rank-sum test.
  The proportion of tumor shrinkage will be examined at visit 7. The between-group differences were examined by McNemar test

SECONDARY OUTCOMES:
Progression-free survival, Largest diameter of tumor, estimated tumor volume | 48th week
  The secondary objective is to assess the effect of cabergoline via measurement of progression -free survival (PFS) over the 48 week-treatment period.

OTHER OUTCOMES:
The change of tumor diameter (mm) | Baseline, 48th week
  The largest diameter (mm) of tumor will also be recorded and compared between groups.
The change of tumor volume (mm³) | Baseline, 48th weeks
  The estimated volume of tumor ( mm³) will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No